CLINICAL TRIAL: NCT04800003
Title: The Gonial Angle as a Predictive Marker of Mandibular Fossa Depth on Panoramic Radiographs: A Diagnostic Accuracy Study
Brief Title: The Gonial Angle as a Predictive Marker of Mandibular Fossa Depth
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Poyzan Bozkurt, Associate Professor, Ankara University
Other Study IDs: 13/1
Record Dates: First submitted 2021-03-15; First posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Dental Implants; Submandibular Fossa Depth; Gonial Angle; Cone-beam Computed Tomography; Panoramic Radiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dry human mandibles, selected for evaluation: 51 dry mandibles with posterior region endetulism and sufficient bone integrity to make the necessary measurements were evaluated. CBCT images of the 51 dry human mandibles included in the study were obtained using the Planmeca Promex-3D (Helsinki, Finland) device in our faculty Dentomaxillofacial Radiology department. Gonial angle was measured on CBCT images as the angle between the tangent line drawn posterior to the border of the ramus of the mandible and the tangent line drawn to the lower border of the mandible. While determining the depth of the submandibular fossa, a line was drawn to connect the most dislocated upper and lower points on the inner surface of the mandible in the coronal plane sections obtained with CBCT, and the length of the line drawn at a right angle from the deepest point of the fossa to this line was measured as the depth of the submandibular fossa.
  Interventions: Diagnostic Test: Gonial angle and submandibular fossa depth measurements from CBCT images

INTERVENTIONS:
Diagnostic Test: Gonial angle and submandibular fossa depth measurements from CBCT images — CBCT images were obtained from dry human mandibles

SUMMARY:
The aim of the study is to evaluate the relationship between submandibular fossa depth and gonial angle measurements in cone beam computed tomography examinations in terms of dental implant applications. Cone-beam computed tomography images of 51 dry human mandibles were included in the study.

DETAILED DESCRIPTION:
Gonial angle and fossa depths were determined and evaluated separately for left and right sides. Gonial angle was measured on Cone-beam computed tomography images as the angle between the tangent line drawn posterior to the border of the ramus of the mandible and the tangent line drawn to the lower border of the mandible. Determination of the submandibular fossa depth was made with a line was drawn to connect the most dislocated upper and lower points on the inner surface of the mandible in the coronal plane sections, and the length of the line drawn at a right angle from the deepest point of the fossa to this line. Measurements were made separately for left and right sides.

ELIGIBILITY:
Inclusion Criteria:

* Dry mandibles with sufficient bone integrity to make the necessary measurements

Exclusion Criteria:

* Dry mandibles which were dentate in the posterior region

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: In the present diagnostic accuracy study, 75 dry human mandibles were used. 24 dry human mandibles with insufficient bone integrity to make the necessary measurements or which were dentate in the posterior region were not included in the study and the study was carried out with 51 dry mandibles.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Gonial angle | 2 months
  Gonial angle and fossa depths were determined and evaluated separately for left and right sides. Gonial angle was measured on CBCT images as the angle between the tangent line drawn posterior to the border of the ramus of the mandible and the tangent line drawn to the lower border of the mandible.
Submandibular fossa depth | 2 months
  A line was drawn to connect the most dislocated upper and lower points on the inner surface of the mandible in the coronal plane sections obtained with CBCT, and the length of the line drawn at a right angle from the deepest point of the fossa to this line was measured as the depth of the submandibular fossa. These measurements were noted as 'millimeters' separately for left and right sides.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No